CLINICAL TRIAL: NCT07086950
Title: Neurorehabilitation of Cognitive Deficits in Multiple Sclerosis Using an Adaptive Cognitive Exergame - Randomized, Controlled, Multi-center Clinical Trial
Acronym: REALISE-MS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Prof. Arseny Sokolov, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Prof. Arseny Sokolov, MD, PhD, Chair and Full Professor of Neurorehabilitation, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REALISE-MS
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Neurorehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Brain Trainer software (Experimental)
  Interventions: Device: Body Brain Trainer software
- RehaCom software (Active Comparator)
  Interventions: Device: RehaCom software

INTERVENTIONS:
Device: Body Brain Trainer software — Patients will engage in cognitive and physical exercises with the training software Body Brain Training (BBT) for 4 consecutive weeks. Participants will be asked to complete 3 sessions per week for a length of ~1h per session.
  Arms: Body Brain Trainer software
Device: RehaCom software — Patients will engage in exercises with the cognitive training software RehaCom (Hasomed®), which is a proxy to the standard of care, for 4 consecutive weeks. Participants will be asked to complete 3 sessions per week for a length of ~1h per session.
  Arms: RehaCom software

SUMMARY:
Approximately 2.8 million people worldwide suffer from multiple sclerosis (MS). In 40 to 70% of cases, individuals with MS experience cognitive impairments that significantly interfere with their personal lives, careers, and quality of life. Current pharmacological and neurorehabilitation treatment options do not adequately reduce cognitive deficits. The absence of standards of care in Switzerland or internationally regarding cognitive neurorehabilitation in MS highlights the need for effective interventions with lasting effects.

To address this need, we are exploring different approaches to support and improve cognitive impairments through training exercises using computerized tools. Traditionally, these exercises are in paper-and-pencil format, consisting of tests, puzzles, and memory tasks. While this approach is useful, computerized tools now allow us to offer more playful, interactive, and engaging approaches.

In this study, we are examining the effect of serious video games (a medical device) on cognitive deficits related to MS. The serious video games we are testing have already been evaluated at CHUV in individuals with MS and cognitive impairments. This recent study demonstrated the feasibility and safety of using these games in people with MS. With the current study, we aim to test these tools on a larger scale in order to better understand their effects on cognitive functions. More specifically, we seek to determine which of the two proposed interventions provides the greatest cognitive benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent signed by the participant,
2. Adults 18+ years,
3. Patients with a diagnosis of relapsing multiple sclerosis according to the most recent internationally recognized criteria, as evaluated by their treating physicians (Thompson et al., 2018) or secondary progressive MS (diagnosis ≤ 30 months),
4. Presence of cognitive complaint,
5. Z-Score ≤ -0.5 in the Symbol Digit Modalities Test (SDMT)

Exclusion criteria:

1. Clinically or radiologically confirmed MS relapses within 3 months prior to enrollment,
2. Change in disease modifying treatments (DMT), antidepressant or anxiolytic medication within 1 month prior to enrollment,
3. High risk of falls based on a completion time of more than 15 seconds in the Four Square Step Test (FSST) (Dite & Temple, 2002),
4. Assisted locomotion or falls in the past 3 months as evaluated in the enrollment interview (Hopkins Falls Grading Scale (Grade > 1)),
5. Major psychiatric and/or neurocognitive disorders according to the DSM-5 (APA, 2013),
6. Incapacity to discriminate colors (Ishihara test; (Clark, 1924)),
7. Insufficient language knowledge to understand instructions or questionnaires,
8. High-risk pregnancy as evaluated by the appointed gynecologist.
9. Z-Score ≤ -3.5 in the Symbol Digit Modalities Test (SDMT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
PDQ-20 | End of training period (4 weeks).
  The primary endpoint of this clinical trial is the change in subjective cognitive dysfunction, as measured by the Perceived Deficits Questionnaire-20 (PDQ-20) total score, in people with multiple sclerosis using exergame (BBT) compared to RehaCom (control) from baseline to end-of-training.

IPD SHARING:
Plan to Share IPD: Yes